CLINICAL TRIAL: NCT06020950
Title: Effects of Chia Seed Consumption in Comparison With Marine Omega-3 Supplementation on the Concentration of Blood Lipid and Inflammatory Factors in Hypertriglyceridemic Patients
Brief Title: Chia Seeds Consumption in Hypertriglyceridemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 43005340
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Salvia hispanica seed extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Reduced calorie diet along with placebo (sunflower oil) pearls
  Interventions: Other: Control
- Omega-3 supplementation (Active Comparator): Reduced calorie diet along with omega-3 supplementation
  Interventions: Dietary Supplement: Omega-3 supplementation
- Chia seed (Experimental): Reduced calorie diet along with chia seed consumption
  Interventions: Other: Chia seed

INTERVENTIONS:
Other: Control — Low-calorie diet with the use of placebo pearls (containing sunflower oil)
  Arms: Control
Dietary Supplement: Omega-3 supplementation — Low-calorie diet with the use of marine omega-3 pearls (containing 1200 mg eicosapentaenoic acid + 600 mg docosahexaenoic acid/day)
  Arms: Omega-3 supplementation
Other: Chia seed — Low-calorie diet with the consumption of 30 grams of powdered chia seeds
  Arms: Chia seed

SUMMARY:
Lifestyle changes including diet therapy and weight loss can improve hypertriglyceridemia (HTG) . Furthermore, increasing omega-3 fatty acids intake has therapeutic effects on HTG. Alpha-linolenic acid is the precursor of long-chain omega-3 fatty acid and it is abundant in sources such as chia seeds and flax seeds. Considering the high fiber and omega-3 content of chia seeds and the existing mechanisms for improving lipid profile through fiber and omega-3, animal studies have shown the positive role of chia seed consumption on lipid profile, glycemic and lipid factors, and inflammation. However, in human studies, conflicting results have been obtained and some studies have shown beneficial effects on blood lipid, glycemic, and inflammatory factors, but in some studies, no effect has been observed. The objective of this study is to determine the effects of chia seed consumption on lipids, glycemic and inflammatory factors in people with HTG.

DETAILED DESCRIPTION:
This study is an unblinded randomized controlled clinical trial. The study will be conducted on people with mild to moderate hypertriglyceridemia whose fasting blood triglyceride levels were between 150-499 mg/dL in the previous two tests. Participants who meet the following criteria will not be included in the study: Being treated with fibrate medications, end-stage kidney disease, acquired immunodeficiency syndrome patients, cancer patients undergoing chemotherapy or radiotherapy, patients with liver cirrhosis, being treated glucocorticoids, continuous use of omega-3 supplements or in the past month, and pregnancy or lactation.

Patients will be randomly assigned to one of three study groups. The duration of the study will be 8 week. The groups are: the control group, which is given a placebo pearls containing sunflower oil. the omega-3 oil group will be given omega-3 pearls, and the chia seed group that will consume chia seeds. In addition, the participants of all three groups are subjected to a low-calorie diet. At the beginning and end of the study, the measurements include body weight, blood pressure, blood concentration of lipids, lipoproteins and inflammatory factors.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals who had fasting triglyceride concentration 150-499 mg/dL in their two previous tests

Exclusion Criteria:

* Being treated with fibrate medications
* Being treated glucocorticoids
* Being treated with anticoagulants (except aspirin)
* Continuous use of omega-3 supplements or in the past month
* End-stage kidney disease
* Acquired immunodeficiency syndrome patients
* Cancer patients undergoing chemotherapy or radiotherapy
* Patients with liver cirrhosis
* Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of triglycerides | 8 week
  Fasting plasma concentration of C-reactive protein and IL-6

SECONDARY OUTCOMES:
Weight loss | 8 week
  Body wight loss (kg)
Plasma concentration of insulin | 8 weeks
  Fasting plasma concentration of insulin
Plasma inflammatory factors concentration | 8 week
  Fasting plasma concentration of C-reactive protein and IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Unit, National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shahparvari MR, Nasrollahzadeh J. Effect of chia seeds or concentrated fish oil on cardiometabolic risk markers in subjects with hypertriglyceridaemia: a parallel clinical trial. J Hum Nutr Diet. 2024 Dec;37(6):1558-1570. doi: 10.1111/jhn.13369. Epub 2024 Oct 3. PMID 39360590